CLINICAL TRIAL: NCT04519021
Title: Knowledge, Attitude and Practice Regarding Diagnosis and Management of Gout Among Clinicians in Nepal: A Report From Web-Based Survey
Brief Title: Knowledge, Attitude and Practice Regarding Diagnosis and Management of Gout Among Clinicians in Nepal
Status: Completed | Type: Observational
Sponsor: National Center for Rheumatic Diseases, Nepal (Other)
Responsible Party: Sponsor
Other Study IDs: 07/2076
Record Dates: First submitted 2020-08-16; First posted 2020-08-19 (Actual); Last update posted 2020-08-19 (Actual); Status verified 2020-08

CONDITIONS: Gout
Keywords: gout; survey; knowledge; practice; nepal
MeSH Terms: conditions — Gout

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
A web-based descriptive survey was conducted among doctors with regular interaction with gout patients. The questionnaire comprised of 38 multiple choice questions; 9 questions for demographic data, 8, 11 and 10 questions each for knowledge, attitude and practice, respectively. Simple descriptive statistics were used to describe the correct responses.

DETAILED DESCRIPTION:
Objective To understand the knowledge, attitude and treatment practices of gout among doctors who regularly interacted with gout patients.

Methodology Study population: Physicians (including practicing medical graduates, post-graduates in internal medicine, family medicine) and orthopedic surgeons were selected randomly from the list of data from the Nepal Medical Council registry. All internists with valid email ID on the registry of the "society of internal medicine of Nepal" (SIMON) were included. Also, a list of MBBS graduates, family medicine and orthopedic practitioners working in the peripheral set-up of Nepal was obtained and a random selection with computer-generated random number table based on council registration number was made for enrollment into the survey. Estimating a response rate of 30%, a total of 1200 clinicians were selected based on their council registration number for the invitation to participate in the survey.

Survey instrument: A standardized questionnaire was designed by a 3-member committee of NRA focusing on the areas of knowledge, attitude and practice of gout with 9 questions pertaining to demographic parameters, 8 to knowledge about the disease, 11 to attitude and 10 to practice behaviors [tables 1-4]. The questions were designed as multiple-choice questions (MCQ) to be marked by the respondent. Few questions had the provision of selecting more than 1 options. Open- ended questions were avoided to save the time of the respondents and thus reduce the attrition rates[10].

Procedure: An email containing a letter of invitation for participation was sent to each of the selected participant. It mentioned why they were receiving the email, the objectives of the survey, the assurance of anonymity and confidentiality and a total answering time of less than 5 minutes for encouraging participation. A link to the Google-form was attached in the mail itself and a mention was made on the implied consent for participation in clicking the link. A reminder email was sent after 1 week to all irrespective of whether they had responded earlier.

Platform: A web-based platform was chosen with the use of Google-forms which was compatible and user friendly to both browser and mobile users and to both iOS and Android users. Multiple entries from the same email link were blocked. Web-based platform was chosen over email survey because it provides the ability to transfer survey responses directly into a database, eliminating transcription errors and preventing survey alteration by the survey respondent and most importantly maintaining confidentiality and anonymity of respondents[11]. The answers were collected anonymously in an excel sheet at the main server for analysis.

Statistical analysis: Simple descriptive statistics were used to describe the frequency or correct responses. Chi-square test was performed to assess the difference in knowledge, attitude, and practices between clinicians with different medical qualifications. Analysis was done using SPSS version 21 (SPSS, Inc., Chicago, IL, USA).

ELIGIBILITY:
Inclusion Criteria:

* Physicians (including practicing medical graduates, post-graduates in internal medicine, family medicine)
* orthopedic surgeons
* with valid email ID on the registry of the "society of internal medicine of Nepal" (SIMON)

Exclusion Criteria:

* who did not give consent
* clinicians other than above mentioned faculty

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Physicians (including practicing medical graduates, post-graduates in internal medicine, family medicine) and orthopedic surgeons were selected randomly from the list of data from the Nepal Medical Council registry. All internists with valid email ID on the registry of the "society of internal medicine of Nepal" (SIMON) were included.
Sampling Method: Non-Probability Sample
Enrollment: 380 (Actual)
Dates: Start 2019-11-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2020-01-31 (Actual)

PRIMARY OUTCOMES:
evaluation of knowledge | 3 months
  evaluation of knowledge on gout among clinicians
evaluation of attitude | 3 months
  evaluation of attitude on gout among clinicians
evaluation of practice | 3 months
  evaluation of practice on gout among clinicians

CONTACTS AND LOCATIONS:
Locations (1):
- National center for Rheumatic Diseases, Kathmandu, Nepal

IPD SHARING:
Plan to Share IPD: Undecided